CLINICAL TRIAL: NCT04485429
Title: Efficacy Assessment of Methylprednisolone and Heparin in Patients With COVID-19 Pneumonia: A Randomized, Controlled, 2x2 Factorial Study
Brief Title: Efficacy Assessment of Methylprednisolone and Heparin in Patients With COVID-19 Pneumonia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: It was not possible to perform the study due to the availability and logistics of porcine heparin
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 31180820600005249
Record Dates: First submitted 2020-07-20; First posted 2020-07-24 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Heparin; Methylprednisolone; Anticoagulation; Coagulopathy; Respiratory failure
MeSH Terms: conditions — COVID-19; Hemostatic Disorders; Respiratory Insufficiency | interventions — Methylprednisolone; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Methylprednisolone + Standard treatment (Experimental): Participants will receive the standard treatment and methylprednisolone.
  Interventions: Drug: Methylprednisolone
- Full-dose heparin + Standard treatment (Experimental): Participants will receive the standard treatment and full-dose heparin,
  Interventions: Drug: Heparin
- Methylprednisolone + Full-dose heparin + Standard treatment (Experimental): Participants will receive the standard treatment, methylprednisolone and full-dose heparin
  Interventions: Drug: Methylprednisolone; Drug: Heparin
- Standard treatment (No Intervention): Participants will receive the standard treatment

INTERVENTIONS:
Drug: Methylprednisolone — Methylprednisolone 0.5 mg/kg every 12 hours intravenously for the first 14 days; followed by 0.5 mg/kg/day from day 15 to day 21; followed by 0.25mg/kg/day from day 22 to day 25; followed by 0.125 mg/kg/day, from day 26 to day 28 of treatment.
  Arms: Methylprednisolone + Full-dose heparin + Standard treatment; Methylprednisolone + Standard treatment
Drug: Heparin — Enoxaparin 1 mg/kg subcutaneously every 12 hours (if creatinine clearance greater than 40ml/min) or Unfractionated heparin dosed to target activated partial thromboplastin time (aPTT) between 1.5 - 2.0 times the normal value (if creatinine clearance less or equal to 40ml/min). The treatment period with full-dose heparin will be 7 days. After 7 days of full-dose heparin, patients will continue using prophylactic dose of heparin, according to the standard treatment routine.
  Arms: Full-dose heparin + Standard treatment; Methylprednisolone + Full-dose heparin + Standard treatment

SUMMARY:
The COVID-19 pandemic has been spreading continuously, and in Brazil, until July 19, 2020, there have been more than 2,000,000 cases with more than 79,000 deaths, with daily increases. The present study proposes to evaluate the efficacy of methylprednisolone and heparin in treatment of patients with COVID-19 pneumonia in a randomized, controlled, 2x2 factorial study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 by RT-PCR or serology with presence of IgM positive antibodies;
* Lung image (X-ray or chest CT) with involvement of at least 25% of the parenchyma;
* O2 saturation in ambient air less than or equal to 93%
* Alteration of inflammatory tests

  * D-Dimer above the reference value and
  * Elevation of C-reactive protein, ferritin or lactic dehydrogenase
* Sign the consent form.

Exclusion Criteria:

* QT interval prolongation
* Imminence of orotracheal intubation (intubation prediction in the first 4 hours after randomization)
* Women who are pregnant or breastfeeding
* Corticosteroid allergy or intolerance
* Chronic corticosteroid users (prednisone equivalent > 10 mg daily)
* Patients diagnosed with cancer with increased bleeding potential
* Patients in hemodialysis
* History of peptic ulcer
* Herpes zoster infection
* History or active treatment of tuberculosis
* Systemic fungal infection
* Use of anticoagulation due to previous pathology
* Glaucoma
* Live virus vaccine up to 90 days before randomization
* Known coagulopathy or thrombocytopenia (<40,000/mm3) or hypofibrinogenemia (< 50 mg/dL)
* Recent bleeding
* Another limiting comorbidity for administering the therapies provided for in this protocol in in researcher's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of invasive mechanical ventilation | 28 days

SECONDARY OUTCOMES:
Severity assessment by ordinal severity scale | 3 days, 7 days, 14 days, 28 days after randomization
  Severity assessment will be performed using the ordinal severity scale during hospitalization.
Severity assessment by SOFA score | 3 days, 7 days, 14 days, 28 days after randomization
  Severity assessment will be performed using the SOFA score during hospitalization.
Length of hospital stay | 28 days
Length of stay in intensive care | 28 days
Death rate | 14 days, 28 days, 60 days, 90 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M Rego, MD, PhD, Principal Investigator — D'Or Institute for Research and Education
Locations (1):
- D'Or Institute for Research and Education, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208